CLINICAL TRIAL: NCT05269797
Title: The Implementation and Initial Impact of a Nurse-led Health Coaching Intervention for Heart Failure Self-care Management
Brief Title: A Nurse-led Health Coaching Intervention for Heart Failure Self-care Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Victoria Smye
Record Dates: First submitted 2022-01-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Behavioural
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health-coaching Intervention (Experimental): A nurse-lead health coaching intervention to support heart failure self-care management is employed by the nurses. This is a pre-post single group design - there is only one arm.
  Interventions: Behavioral: Nurse-led health coaching re: heart failure self-care management

INTERVENTIONS:
Behavioral: Nurse-led health coaching re: heart failure self-care management — A focus group meeting will be arranged with the nurse participants to provide training on the study intervention specific to the Nurse-led health coaching intervention. The intervention involves identifying barriers and finding strategies and solutions to self-care management, while employing a self-care HF management tool of adjusting diuretic dosing (ADD) according to the congestive cardiac calendar (designed in collaboration with nurses in Phase 1). It will be essential for the nurses to document key information pertaining to the rationale for these decision-making strategies or solutions. This is in comparison to the standard of care in primary health care of nurses not taking a standardize approach towards health coaching and the patient being instructed by the practitioner to take a set diuretic dosing (SDD).

SUMMARY:
There is an increase in Heart Failure (HF) hospitalizations and readmissions despite medical advances (Desai & Stevenson, 2012; Ambrosy et al.,2014) and in spite of the education provided to HF patients regarding the signs of fluid accumulation, HF exacerbations persist. Unfortunately, there seems to be a gap between patients recognizing these signs of fluid accumulation and performing timely self-management activities to control it. Currently, there is no standardized approach for the delivery of a nurse-led health coaching intervention to assist patients to engage in HF symptom management with self-care activities within a Primary Health Care (PHC) setting. To address this gap, the aim of this research is to examine the feasibility, acceptability, and initial effectiveness of a nurse-led health coaching intervention, involving a self-care activity of the Adjusted Diuretic Dosing (ADD) tool with stable HF patients and their significant others a PHC approach and within a PHC setting.

In the proposed study, nurses will engage with health coaching and a health coaching tool (developed in Phase 1 of this research with the assistance of nurses working in this area) to assist the patient to identify barriers to self-care and develop the patient's goals to successfully engage in HF self-care strategies. It is also necessary for the nurse to capture through documentation what decision-making strategies the nurse performed to assist the patient with HF management. It is through these decision-making points, identified strategies can be examined by the researcher to determine what care gaps or process has occurred. Also, It is through the awareness of the patient's knowledge, skills, past experience, and values and beliefs, those daily decisions will be made by the patient, e.g., decisions will be influenced by the interactions among the person, the problem, and setting or environment - they are situation-specific (Riegel et al., 2016). It is expected that through this kind of naturalistic decision-making process the patient's self-confidence will increase to take action towards maintaining HF self-care activities (such as medication and diet adherence, and weight monitoring), respond to the perception of HF symptoms (seeking medical attention), and be supported to manage their HF condition (adjusting diuretics in response to fluid retention); this to support improved health outcomes and quality of life.

DETAILED DESCRIPTION:
Purpose of the Study:

To determine the feasibility and acceptability of a nurse-led health coaching intervention to support heart failure self-care management.

Hypothesis: A nurse-led health coaching intervention will engage patients to take action in self-care activities that have the potential to increase self-care confidence and quality of life for both the patient and their caregiver that will be measured by the Minnesota Living with HF Questionnaire (MLHFQ) and Self-Care HF Index (SCHFI), and Caregiver Contribution for Self-Care HF Index (CC-SCHFI).

It is an expectation the results of this study will inform nursing practice in this domain; the results from this research study have the potential to improve the quality and consistency of HF patient care with improved outcomes for persons living with HF.

Qualitative Research Questions:

1. What are those key elements of the nurse-led health coaching intervention that facilitated or challenged the nurses' experiences to implement HF self-care management? (nurse consultants in a focus group format)?
2. What are those elements of the nurse-led health coaching intervention that were helpful and/or hindered patient experiences of self-management? (Feasibility: A focus group interview with nurses and individual in-depth interviews with patient/caregiver dyads).
3. What is the impact of a nurse-led health coaching intervention? (A focus group interview with nurses and individual in-depth interviews with patient/caregiver dyads).

This is a prospective, non-randomized, single dyad group cohort study utilizing purposive sampling to enroll 6 -10 patients with HF and their caregivers (i.e., 6-10 dyads) over a period of 6 months. The study design type will be conducted as a pre-post pilot feasibility study since the primary objective is to evaluate the feasibility, acceptability, and effectiveness of the health coaching intervention involving a self-care activity of the Adjusted diuretic dosing (ADD) tool with stable HF for patients and their significant others (through qualitative interviews with patients/spouses and nurses) in a family health care setting. This study also will incorporate qualitative methods informed by interpretive description to understand the experiences and decision-making strategies of the nurse employing the intervention and the patient/caregiver dyad engaging in the intervention, i.e., in-depth nurse focus group and individual (dyad) interviews will be conducted. Identifying what features facilitate nurse health coaching and/or challenge its implementation and those features of nurse-led health coaching that were helpful and/or hindered the patient experience of self-management will inform nursing practice in this realm. The secondary objectives are related to evaluating 'trends' (due to an underpowered study) in specific pre-post outcomes associated with the intervention. These identified trends involving characteristics of Quality of Life (QoL) and self-care confidence will be measured by the Minnesota Living with HF Questionnaire (MLHFQ) and Self-Care HF Index (SCHFI), and Caregiver Contribution for Self-Care HF Index (CC-SCHFI) will provide a deeper understanding of the qualitative data.

Patient population procedures:

Heart failure (HF) patients' standard of care can include frequent clinic visits from weekly to every three months depending if HF medication therapy has been initiated or adjusted (i.e., diuretics or ace-inhibitors). Also, it may include routine laboratory blood tests to monitor electrolytes, renal function, and complete blood count. Other possible diagnostic investigations that may be ordered as part of routine care according to evidence-based HF guidelines include an echocardiogram, electrocardiogram, or chest x-ray.

In regard to the care management within a PHC setting, currently, nurses are not leading to take a standardized approach towards health coaching and the practitioner prescribes a set diuretic dosing (i.e., Lasix 40mg p.o. daily) with no opportunity to health coach on self-adjust diuretic if HF symptoms worsen and weight gain has occurred. For this study, an analysis of a nurse leading a health coaching approach by implementing the intervention to identify challenges or barriers to HF self-care management and identifying strategies or solutions with the patient and their caregiver will be conducted. Support from the care team practitioners, either a Nurse Practitioner or family physician will be responsible and lead medication adjustments by prescribing an adjusted diuretic dosing (ADD) which is the self-care management tool within the health coaching intervention (i.e., baseline Lasix 40mg daily, adjust Lasix 40 mg twice a day if weight gain of 3 lbs or more a day).

Nurse-led intervention:

A nurse-led health coaching HF self-care management intervention that is protocol-specific to this study will be implemented. This involves a nurse leading a health coaching approach by implementing the intervention with the patient to identify challenges or barriers to HF self-care management and identifying strategies or solutions. This will be carried out at baseline, 1 and 3-month clinic visits & during the phone visits @ 2 weeks and 8 weeks. If the patient's symptoms deteriorate in between scheduled study visits, the patient will be instructed at the start of the study that they need to contact the clinic to be seen by either the Nurse Practitioner or physician as per current clinic practice and standard of care. This clinic visit details will be documented in the electronic medical record (EMR) and will be captured in the study as a non-schedule visit for the study by the study nurse participant. The patient is also expected to weigh themselves every morning and record it, along with any symptoms they may be experiencing on the "Cardiac congestion calendar" which is part of the intervention that is provided to the patient.

The patient will complete a self-care confidence survey SCHFI (Self-care heart failure index) and a quality-of-life questionnaire MLHFQ (Minnesota living heart failure questionnaire) at the initial visit (baseline) and at the end of the study. The patient will be interviewed separately via audio at the end of the study to explore their self-care management experiences. This can be done either in the clinic or by phone.

ELIGIBILITY:
Inclusion criteria: Patient

* Adult HF patients (age 18 years or older) with a documented diagnosis of HF on the medical record who are stable with no acute signs of HF decompensation and on a stable dose of diuretics for a minimum of three months.
* Patients registered within the Family Medical Clinics in London who have a caregiver or support defined by a person who provides either direct HF support (medication or meal preparation) or indirect HF support (providing emotional support, transportation, or assisting with decision-making around symptom perception or management).
* Patient and caregiver dyads who have a willingness and ability to participate in an interview and complete surveys; and
* English speaking.

Inclusion Criteria: Nurses

-Registered nurses, including Nurse Practitioners employed at the Family Medical Clinics in London who participate in the care of patients living with HF.

Exclusion Criteria: Patients

* A person with cognitive impairment that would interfere with their ability to provide informed consent.
* A person with any medical condition that has an expected survival of less than 6 months: End-stage renal disease, end-stage liver disease, end stage Chronic Obstructive Pulmonary Disease (COPD), end-stage/terminal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale on the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Baseline
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a 21-item paper self- administered questionnaire designed as a measure of heart failure, as indicated by its adverse effects on patients' lives. The MLHFQ quantifies a single overall score as a measure of the impact of heart failure on the patient's life. Higher scores indicate worse physical and emotional quality of life. Physical 0-40 Emotional 0-25
Patient Self Confidence on the Self-Care Heart Failure Index (SCHFI) | Baseline
  Patient Self-Confidence on the Self-Care Heart Failure Index (SCHFI) measures self-care with three scales: self-care maintenance, measuring behaviors to maintain HF stability; symptom perception, measuring monitoring behaviors; and self-care management, assessing the response to symptoms.Physical 0-40 Emotional 0-25 Scores 0-100.
Caregiver Self Confidence on the Caregiver Contribution for Self-Care Heart Failure Index (CC-SCHFI) | Baseline
  The Caregiver Contribution to Self-Care of Heart Failure Index (CC-SCHFI) measures these contributions across three scales: self-care maintenance (symptom monitoring and treatment adherence); self-care management (dealing with symptoms); and confidence in contributing to the self-care (self-efficacy in managing self-care). Higher scores indicating greater caregiver contributions to heart failure self-care. Scores 0-100.

SECONDARY OUTCOMES:
Changes in the Quality of Life Scale on the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 6 months
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a 21-item paper self- administered questionnaire designed as a measure of heart failure, as indicated by its adverse effects on patients' lives. The MLHFQ quantifies a single overall score as a measure of the impact of heart failure on the patient's life. Higher scores indicate worse physical and emotional quality of life; Physical 0-40, Emotional 0-25.
Changes in Patient Self Confidence on the Self-Care Heart Failure Index (SCHFI) | 6 months
  Patient Self-Confidence on the Self-Care Heart Failure Index (SCHFI) measures self-care with three scales: self-care maintenance, measuring behaviors to maintain HF stability; symptom perception, measuring monitoring behaviors; and self-care management, assessing the response to symptoms. Higher scores indicating better self-care. Scores 0-100.
Changes in Caregiver Self Confidence on the Caregiver Contribution for Self-Care Heart Failure Index (CC-SCHFI) | 6 months
  Caregiver Contribution for Self-care Heart Failure Index (CC-SCHFI) measures these contributions across three scales: self-care maintenance (symptom monitoring and treatment adherence); self-care management (dealing with symptoms); and confidence in contributing to the self-care (self-efficacy in managing self-care).Higher scores indicating greater caregiver contributions to heart failure self-care. Scores 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Smye, PhD, Principal Investigator — Western University